CLINICAL TRIAL: NCT02308358
Title: Long Term Outcomes of Osteochondral Allografts for Osteochondral Defects of the Knee.
Acronym: LongTermOC
Status: Withdrawn | Type: Observational
Why Stopped: New study initiated to replace this one
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Stannard, Professor and Chairman - Orthopaedic Surgery, University of Missouri-Columbia
Other Study IDs: 1210204
Record Dates: First submitted 2014-11-14; First posted 2014-12-04 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Outcomes of Allograft
Keywords: Osteochondral Defect; Femoral condyle osteochondral defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Allograft Transplantation: Subjects with femoral condyle osteochondral defects ≥10mm, as determined by MRI or diagnostic knee arthroscopy, will be recruited for allograft transplantation.
- Microfracture Treatment: Subjects with femoral condyle osteochondral defects <10mm, as determined by MRI or diagnostic knee arthroscopy, will be recruited for microfracture treatment.

SUMMARY:
The purpose of this study is to evaluate the functional and clinical outcomes of patients receiving femoral condyle osteochondral allografts, to evaluate potential predisposing factors to failure of such grafts, and to compare the overall outcomes of the grafts to the current standard of care for smaller lesions, microfracture. Our hypothesis is that patients treated with these allografts will demonstrate significant functional improvement as measured by validated outcome scoring measures and their function will be at least equal to that of microfracture outcomes.

DETAILED DESCRIPTION:
Localized articular cartilage defects are a common and challenging problem, particularly in young patients. These defects cause significant disability and, as participation in sports activity grows, are increasing in overall number annually. A recent systematic review evaluating the overall full-thickness focal chondral defects in athletes revealed the prevalence to be 36%, with 22% of the athletes being symptomatic. As the prevalence of these injuries increases, they pose increasingly significant challenges to the clinicians who treat them.

Normal joint cartilage is a firm, elastic tissue that covers the ends of bones to protect them and allow smooth, pain-free movement over each other. Joint cartilage is described, macroscopically and microscopically, as articular or "hyaline" cartilage. Hyaline cartilage is often described as a "glass-like" structural tissue because of its shiny appearance and translucency. The tissue structure is a hydrated matrix consisting of proteoglycans and at least 90% (dry weight) Type II collagen fibers. The collagen fibers contribute to the overall tensile strength and the proteoglycans provide the stiffness and tissue resiliency. Cartilage cells, or chondrocytes, produce dense matrix, which effectively incarcerate the cells themselves. In the event of injury, the motility of these cells is restricted due to their inclusion deep inside the matrix, and the avascularity of the cartilage itself. This lack of a vascular network prevents the infiltration of inflammatory cells and bioactive molecules following damage. Thus, once damaged, adult articular cartilage will not effectively heal or regenerate.

Treatment techniques of osteochondral lesions are relatively new and frequently changing and evolving. The treatment algorithms for these injuries are complex and often involve multiple procedures, including non-surgical interventions with pharmacological agents such as oral non-steroidal anti-inflammatory drugs (NSAIDs), injectable corticosteroids, and activity modification including rehabilitation and support braces that may provide incomplete or temporary relief. Lesion characteristics such as grade and thickness may also impact treatment options and recovery. Arthroscopic debridement and lavage is effective as a first-line surgical approach for subjects with low physical demands. This procedure eliminates debris and decreases inflammation in the joints, but the symptomatic relief is usually transient and the lesion is not repaired. Treatments providing long-term results may be achieved through a variety of surgical options.

There are many surgical treatments options currently available and each have limitations. Marrow stimulation techniques include microfracture, drilling, and abrasion arthroplasty. The Microfracture technique has been described to address lesions up to 1 cm2 while other authors cite more specific applications depending on lesion size, patient age and physical demands. While microfracture is considered a reparative treatment, the procedure can produce less than optimal results because of the inferior nature of fibrocartilaginous tissue formed. Unlike the Type II collagen normally found in articular cartilage, fibrocartilage consists predominately of Type I collagen. Because it lacks the long-term wear characteristics of normal hyaline cartilage, fibrocartilage can degrade with time.

ACI is a two-staged procedure developed to treat cartilage defects in the knee. For ACI, a primary arthroscopic procedure is performed to assess the defect and a small amount (200mg to 400 mg) of healthy, autologous cartilage is harvested. The tissue is then expanded using a cell-culture process over a period of several weeks. The expanded cells are then implanted into the area of the defect during a second surgical procedure. Studies have demonstrated through histology and quantitative measurements that ACI produces a "hyaline-like cartilage" with a collagen type II content of between 35 percent and 55 percent. Literature indicates that hyaline cartilage may have greater biomechanical strength and integrity than the fibrocartilaginous tissue generated in lesions treated with microfracture. There are several disadvantages using ACI, however, such as the need for two surgeries. It has increased surgical time due to and it is associated with substantial cost to account for ex vivo cell expansion. Potential postoperative complications related to the periosteal patch include cell leakage, hypertrophy and/or delamination, and unequal chondrocyte distribution within the lesion.

Osteochondral grafting, the direct transplantation of an osteochondral autograft or allograft, is the only technique available on the market that transplants intact hyaline cartilage. Fresh osteochondral allografts use active chondrocytes while avoiding donor site morbidity. The grafts are avascular and aneural, meaning they are immunopriveleged and suitable for transplantation. Autograft plugs are typically used to treat small defects (up to 2.5 cm in diameter) due to donor site size limitation. Osteochondral allografts can be harvested up to 35 mm in diameter or an entire compartment can be resurfaced using a shell technique.Clinical outcome of osteochondral autografts has been documented in various studies as good to excellent, particularly in subjects with isolated femoral lesions. A major benefit of osteochondral allografts is their ability to provide the surgeon with the capability to treat much larger defects. A major drawback of many of the aforementioned treatment options (microfracture, ACI, osteochondral autograft) is their inability to treat such large lesions. Additionally, fresh OCA longevity after implantation has been documented to be as long as 25 years, indicating that this procedure can provide long term relief to patients.

The purpose of this study is to evaluate the functional and clinical outcomes of patients receiving femoral condyle osteochondral allografts, to evaluate potential predisposing factors to failure of such grafts, and to compare the overall outcomes of the grafts to the current standard of care for smaller lesions, microfracture. Our hypothesis is that patients treated with these allografts will demonstrate significant functional improvement as measured by validated outcome scoring measures and their function will be at least equal to that of microfracture outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age ≥18 years
2. Femoral condyle osteochondral defect ≥10mm as determined by MRI or diagnostic knee arthroscopy for allograft transplantation, defect <10mm for microfracture treatment
3. Must be physically and mentally willing and able to comply with postoperative and routinely scheduled clinical and radiographic evaluations.
4. Must be able and willing to follow a standardized rehabilitation protocol.
5. Must be able to read and understand English or a language for which translated versions of the patient reported questionnaires and Informed consent form are available.
6. Must be able to sign informed consent and must voluntarily sign the Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved subject Informed Consent Form.

Exclusion Criteria:

* 1. Presence of ipsilateral articular fractures, knee ligament injuries or extensor mechanism injuries

  2. Presence of severe soft tissue injuries around the knee that have required or may require skin grafting or flap coverage.

  3. Presence of a previous below knee amputation

  4. Presence of inflammatory systemic arthritis or disease involving the index joint (i.e. gout)

  5. Is a prisoner

  6. Is receiving workman's compensation

  8. Subject is mentally incompetent such that would preclude the subject from providing adequate consent and/or complying with study requirements

  9. Based on a clinical history, physical examination and/or subject presentation, subject has, or is suspected to have, a history of alcohol and/or drug abuse that would preclude subject from providing adequate consent and/or complying with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of orthopaedic surgeons in Columbia, Missouri at the University of Missouri-Columbia Hospital and Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain Level | 1 Year
  Subject outcomes will be assessed through validated outcomes scoring systems, including the International Knee Documentation Committee (IKDC), the SF-36 health survey and the Tegner activity scale. These will be completed by the participants prior to the index procedure and at the 3, 6 and 12 month visits and yearly thereafter.
Activity Level | 1 Year
  Subject outcomes will be assessed through validated outcomes scoring systems, including the International Knee Documentation Committee (IKDC), the SF-36 health survey and the Tegner activity scale. These will be completed by the participants prior to the index procedure and at the 3, 6 and 12 month visits and yearly thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: James P Stannard, MD, Principal Investigator — Missouri Orthopaedic Institute; James L Cook, DVM, Study Director — Missouri Orthopaedic Institute
Locations (1):
- University of Missouri-Hospital and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No